CLINICAL TRIAL: NCT00195689
Title: A Multi-Center Continuation Trial for Patients Completing Study M02-518 and M02-570 of the Human Anti-TNF Monoclonal Antibody Adalimumab (D2E7) in Patients With Moderate to Severely Active Psoriatic Arthritis
Brief Title: Safety and Efficacy of Adalimumab in Patients With Moderate to Severely Active Psoriatic Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M02-537
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2007-08-29 (Estimated); Status verified 2007-08

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Human anti-TNF monoclonal antibody/adalimumab

SUMMARY:
The purpose of the study is to assess the long-term safety and clinical efficacy of adalimumab in treatment of moderate to severely active psoriatic arthritis

ELIGIBILITY:
Inclusion Criteria:

* Subject completed study M02-518 or M02-570

Exclusion Criteria:

* Subject prematurely discontinued study M02-518 or M02-570

  * Female subject who is pregnant or breast-feeding or considering becoming pregnant
  * Subject considered by the investigator, for any reason, to be an unsuitable candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2003-08

PRIMARY OUTCOMES:
Safety parameters
ACR 20/50/70
PsARC
HAQ
SF-36
FACTIT Fatigue Scale
Disease progression measurements

SECONDARY OUTCOMES:
Patient reported outcomes
Clinical response indicators

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Paperiello, Study Director — Abbott
Locations (1):
- Global Medical Information-Abbott Laboratories, Abbott Park, Illinois, United States

REFERENCES:
- [Derived] Gladman DD, Mease PJ, Choy EH, Ritchlin CT, Perdok RJ, Sasso EH. Risk factors for radiographic progression in psoriatic arthritis: subanalysis of the randomized controlled trial ADEPT. Arthritis Res Ther. 2010;12(3):R113. doi: 10.1186/ar3049. Epub 2010 Jun 10. PMID 20537151
- [Derived] Mease PJ, Ory P, Sharp JT, Ritchlin CT, Van den Bosch F, Wellborne F, Birbara C, Thomson GT, Perdok RJ, Medich J, Wong RL, Gladman DD. Adalimumab for long-term treatment of psoriatic arthritis: 2-year data from the Adalimumab Effectiveness in Psoriatic Arthritis Trial (ADEPT). Ann Rheum Dis. 2009 May;68(5):702-9. doi: 10.1136/ard.2008.092767. Epub 2008 Aug 6. PMID 18684743